CLINICAL TRIAL: NCT06235463
Title: Effectiveness of the Osteopathic Pedal Pump in Reducing Lower Limb Volume in Older Adults with Chronic Leg Lymphedema
Brief Title: Pedal Pump and Leg Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-2023-254
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Fifty two participants will be randomized to one of two conditions: to receive the osteopathic pedal pump (treatment group) or to receive a light tough treatment (control group).
Who Masked: Investigator
Masking Description: The investigator who will be responsible for carrying out the measurements of lower limb volume via water displacement will be blinded to the condition each participant is randomized to. Withholding this information from the investigator conducing the measurements will prevent this information from influencing how the measurements are conducted and therefore removing bias that could skew the results in support of the study's hypotheses (i.e., that the pedal pump does reduce lower limb volume in older adults with lower extremity lymphedema).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osteopathic Pedal Pump (Experimental): Participant lays supine on the table and the operator stands at foot of table. Operator places hands on the feet, contacting the balls of the feet, and carefully plantar flexing to a slight degree. Operator dorsiflexes the feet to cause the whole body to move cephalad. The body is allowed to rebound back caudad towards foot of the table. The operator times the next dosiflexion motion to occur towards the end of the caudad motion wave. Technique time is 5 minutes.
  Interventions: Other: Osteopathic Pedal Pump
- Light Touch Treatment (Sham Comparator): Participant lays supine on the table and the operator stands at foot of table. Operator places hands on the feet and touches participant body on the balls of the feet, but operator does not palpate feet or lower limbs.
  Interventions: Other: Light Touch Treatment

INTERVENTIONS:
Other: Osteopathic Pedal Pump — Participants randomized to this condition will receive 5 minutes of myofascial release to the thoracic inlet and 5 minutes of the pedal pump technique.
  Arms: Osteopathic Pedal Pump
Other: Light Touch Treatment — Participants randomized to receive the sham treatment will receive light touch from the operator on the base of the neck and the balls of the feet. This light touch is meant to mimic the pedal pump through touching the same areas of the body but without palpating so that no lymphatic fluid is removed from the lower limbs.
  Arms: Light Touch Treatment

SUMMARY:
Chronic lymphedema in the lower extremities is a common problem found in older adults that can result in cellulitis, poor wound healing, venous stasis ulcers, and other comorbidities. Compressive therapies are the present gold standard for the manual treatment of lymphedema in the lower extremities. However, the benefits of these compressive therapies are modest, and they are not well tolerated by older adults. An alternative manual treatment is the osteopathic pedal pump, an osteopathic manipulative treatment, that uses a rhythmical pumping motion instead of compressive force to move interstitial fluid from the lower extremities back to the circulatory system. However, the evidence that the osteopathic pedal pump can reduce volume in the lower extremities remains anecdotal. The aim of this study is to determine if the osteopathic pedal pump can reduce volume in the lower extremities among older adults with chronic lymphedema. Leg volume will be measured using water displacement. Older adults with chronic lymphedema of the lower extremities will be randomly assigned to one of two groups: a treatment group that will receive one session of the osteopathic pedal pump and a control group that will receive one session of a light touch treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years old or older
* Have lower leg lymphedema

Exclusion Criteria:

* Any type of acute medical issue or exacerbation
* A chronic medical condition (e.g., asthma, chronic obstructive pulmonary disease, congestive heart failure)
* An active tissue infection or an open wound in the lower limb
* An active bone fracture
* Acute deep venous thrombosis not fully anticoagulated
* Dementia

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Change in limb volume | The time frame in which the pre and post-treatment measurements will take place in one session that will take approximately 30-45 minutes.
  Difference in lower limb volume, as measured by water displacement, from pre to post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No